CLINICAL TRIAL: NCT05795946
Title: Effects of a Whole Food Based Nutritional Formulation on Trimethylamine N-oxide and Cardiometabolic Endpoints in Healthy Adults.
Brief Title: Standard Process Heart and Gut Health Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Internal changes and unanticipated challenges with recruitment.
Sponsor: Standard Process Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SP0012
Record Dates: First submitted 2023-03-08; First posted 2023-04-03 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Nutrition, Healthy
Keywords: Heart health; B Vitamins; D Vitamins; TMAO; Quality of Life; Healthy Heart

STUDY DESIGN:
Intervention Model Description: 3 groups: 1 for B vitamins only, 1 with B vitamins in addition of D vitamins, and one is diet only.
  This pilot study aims to explore the modulation of TMAO response in healthy adults after supplementation with a whole food matrix-based B vitamins formulation alone, and in combination with vitamin D. The assessments will be compared to the diet only control group.
Who Masked: Participant, Care Provider
Masking Description: The labels for the vitamins will only have the participant ID on them
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Diet Only Group (No Intervention): Diet only: guided diet
- Combination Group (Experimental): Combination of whole food-based B and D vitamins
  Interventions: Dietary Supplement: Whole food-based B and D vitamins
- B Only Group (Experimental): Whole food-based B vitamins
  Interventions: Dietary Supplement: Whole food-based B and D vitamins

INTERVENTIONS:
Dietary Supplement: Whole food-based B and D vitamins — Looking at whole food-based B and D vitamins to reduce TMAO levels and if this can modulate gut diversity
  Arms: B Only Group; Combination Group

SUMMARY:
Standard Process Heart and Gut Health Study

DETAILED DESCRIPTION:
This prospective pilot clinical study will screen 45 healthy participants regularly consuming omnivorous diet (full fat dairy, red meat, eggs, fish) and have elevated serum Trimethyl amine N-oxide (TMAO) levels. Trimethylamine N-oxide (TMAO) is a gut microbiota derived dietary metabolite which is emerging as a significant and independent predictor of cardiovascular disease (CVD) risk mainly through inflammation and oxidative stress pathways. Long term consumption of animal products elevates TMAO levels due to its abundance of TMAO precursors: choline and L-carnitine. As diet plays a key role in altering the microbial composition and subsequent TMAO levels, it is important to investigate if whole food based nutritional formulations can provide the necessary support required to manage TMAO levels and hence, positively impact cardiometabolic endpoints. Towards this end both B and D vitamins have been shown to influence the levels of circulating TMAO while maintaining a healthy gut microenvironment.

This pilot study aims to explore the modulation of TMAO response in healthy adults after supplementation with a whole food matrix-based B vitamins formulation alone, and in combination with vitamin D. The assessments will be compared to the diet only control group.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants (both male and female) aged 25-80 years with omnivorous diet (regular consumption of eggs, red meat, dairy)
* No pre or probiotic consumption during study, no antibiotics during study
* Moderate to high serum levels of TMAO (more than or equal to 4 uM) determined by a standard blood test
* If the participant is on antibiotics, they should finish their medication and wait one month before testing for TMAO as a screening criterion
* Normal blood pressure, non-smokers
* Normal cholesterol
* Participants can communicate and follow instructions
* Participants voluntarily signed and dated an informed consent (ICF), reviewed by an Institutional Review Board (IRB), and provided authorization prior to any participation in the study
* Participants who are willing to take nutritional supplements and have no known food allergies

Exclusion Criteria:

* Vegan and vegetarian participants
* Participants on medically prescribed diet
* Participants not willing to stop consumption of fermented products (plain yogurt, kefir, kombucha, water kefir, miso, pickled vegetables, and sauerkraut) 2 weeks prior to the study start date and during the study timeline as this will interfere with gut microbiome related outcome assessment
* Participants not willing to stop consuming polyphenols- green tea, cocoa, flaxseed, berries, and energy drinks
* Participants who are currently or have participated in other interventional clinical trials in the last 4 weeks
* Participants on certain supplements like GI health related (Probiotics, prebiotics, and/or antimicrobial botanicals), vitamin C, Choline, lecithin or L-carnitine, fish oil/krill oil containing supplements who don't wish to stop supplementation prior to 2 weeks of study start date
* Participants who have any confirmed or suspected infectious disease (such as tuberculosis, Hepatitis B or C, HIV infection), malignancy, or any other clinically significant medical condition, which in the investigators' opinion, makes him or her not suitable for inclusion in the study*
* Participants who have pacemakers, an implanted cardioverter defibrillator (ICD), or a cardiac resynchronization therapy device
* Participants who have confirmed or suspected pregnancy (self-reported)
* Participant waiting for a heart transplant
* Participants currently hospitalized for acute myocardial infarction
* Participants with a planned revascularization within 30 days of screening
* Participants must not have any allergies to supplement ingredients (see list)
* Participants who have initiated the use of prescription medications (defined as a medication that can be prescribed only by a properly authorized/licensed clinician), and not authorized non-prescription medications (over-the-counter medications), and other nutritional supplements
* Participants who do not comply with all study requirements (including clinical visits)
* Participants with high cholesterol or on lipid lowering medications like statins
* Participants on following medication: NSAIDS, Steroids, Prednisone, Acid Reflux/GERD medicines: Tagamet, Zantac, Pepcid, Prilosec, Prevacid

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Primary | 8 weeks
  One outcome is to determine if a combination of whole food-based B-vitamins can modulate gut diversity and TMAO response

SECONDARY OUTCOMES:
Secondary | 8 weeks
  Another outcome is to explore the beneficial interplay between B and D vitamin supplementation in reducing TMAO levels through modulation of gut microbiome.

CONTACTS AND LOCATIONS:
Overall Officials: Chinmayee Panda, PhD, Principal Investigator — Standard Process Inc.
Locations (1):
- Standard Process Nutrition Innovation Center, Kannapolis, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to share data with other researchers

REFERENCES:
- [Background] Kvapil J, Liska M. [Polarimetric determination of D-arabonates]. Cesk Farm. 1965 May;14(4):164-6. No abstract available. Czech. PMID 5837488
- [Background] Ma J, Li H. The Role of Gut Microbiota in Atherosclerosis and Hypertension. Front Pharmacol. 2018 Sep 25;9:1082. doi: 10.3389/fphar.2018.01082. eCollection 2018. PMID 30319417
- [Background] Brunt VE, Gioscia-Ryan RA, Richey JJ, Zigler MC, Cuevas LM, Gonzalez A, Vazquez-Baeza Y, Battson ML, Smithson AT, Gilley AD, Ackermann G, Neilson AP, Weir T, Davy KP, Knight R, Seals DR. Suppression of the gut microbiome ameliorates age-related arterial dysfunction and oxidative stress in mice. J Physiol. 2019 May;597(9):2361-2378. doi: 10.1113/JP277336. Epub 2019 Feb 27. PMID 30714619
- [Background] Sun X, Jiao X, Ma Y, Liu Y, Zhang L, He Y, Chen Y. Trimethylamine N-oxide induces inflammation and endothelial dysfunction in human umbilical vein endothelial cells via activating ROS-TXNIP-NLRP3 inflammasome. Biochem Biophys Res Commun. 2016 Dec 2;481(1-2):63-70. doi: 10.1016/j.bbrc.2016.11.017. Epub 2016 Nov 8. PMID 27833015
- [Background] Zhu W, Wang Z, Tang WHW, Hazen SL. Gut Microbe-Generated Trimethylamine N-Oxide From Dietary Choline Is Prothrombotic in Subjects. Circulation. 2017 Apr 25;135(17):1671-1673. doi: 10.1161/CIRCULATIONAHA.116.025338. No abstract available. PMID 28438808
- [Background] Ketheesan N, Ingham E, Kearney JN, Rasaretnam R. Donor valves as substitutes for heart valve replacement. Ceylon Med J. 1997 Jun;42(2):85-90. PMID 9257469
- [Background] Sohouli MH, Ozovanu OD, Fatahi S, Hekmatdoost A. Impact of probiotic supplementation on trimethylamine N-oxide (TMAO) in humans: A systematic review and meta-analysis of randomized controlled trials. Clin Nutr ESPEN. 2022 Aug;50:56-62. doi: 10.1016/j.clnesp.2022.06.006. Epub 2022 Jun 17. PMID 35871952
- [Background] Wang Q, Guo M, Liu Y, Xu M, Shi L, Li X, Zhao J, Zhang H, Wang G, Chen W. Bifidobacterium breve and Bifidobacterium longum Attenuate Choline-Induced Plasma Trimethylamine N-Oxide Production by Modulating Gut Microbiota in Mice. Nutrients. 2022 Mar 14;14(6):1222. doi: 10.3390/nu14061222. PMID 35334879
- [Background] Dalla Via A, Gargari G, Taverniti V, Rondini G, Velardi I, Gambaro V, Visconti GL, De Vitis V, Gardana C, Ragg E, Pinto A, Riso P, Guglielmetti S. Urinary TMAO Levels Are Associated with the Taxonomic Composition of the Gut Microbiota and with the Choline TMA-Lyase Gene (cutC) Harbored by Enterobacteriaceae. Nutrients. 2019 Dec 25;12(1):62. doi: 10.3390/nu12010062. PMID 31881690
- [Background] Keith ME, Walsh NA, Darling PB, Hanninen SA, Thirugnanam S, Leong-Poi H, Barr A, Sole MJ. B-vitamin deficiency in hospitalized patients with heart failure. J Am Diet Assoc. 2009 Aug;109(8):1406-10. doi: 10.1016/j.jada.2009.05.011. PMID 19631047
- [Background] Zhao LG, Shu XO, Li HL, Gao J, Han LH, Wang J, Fang J, Gao YT, Zheng W, Xiang YB. Prospective cohort studies of dietary vitamin B6 intake and risk of cause-specific mortality. Clin Nutr. 2019 Jun;38(3):1180-1187. doi: 10.1016/j.clnu.2018.04.016. Epub 2018 May 4. PMID 29764693
- [Background] Reay JL, Smith MA, Riby LM. B vitamins and cognitive performance in older adults: review. ISRN Nutr. 2013 Mar 11;2013:650983. doi: 10.5402/2013/650983. eCollection 2013. PMID 24959550
- [Background] Malik M, Hnatkova K, Batchvarov V, Gang Y, Smetana P, Camm AJ. Sample size, power calculations, and their implications for the cost of thorough studies of drug induced QT interval prolongation. Pacing Clin Electrophysiol. 2004 Dec;27(12):1659-69. doi: 10.1111/j.1540-8159.2004.00701.x. PMID 15613131
- [Background] Hsiao PY, Mitchell DC, Coffman DL, Allman RM, Locher JL, Sawyer P, Jensen GL, Hartman TJ. Dietary patterns and diet quality among diverse older adults: the University of Alabama at Birmingham Study of Aging. J Nutr Health Aging. 2013 Jan;17(1):19-25. doi: 10.1007/s12603-012-0082-4. PMID 23299373
- [Background] Borel P, Mekki N, Boirie Y, Partier A, Alexandre-Gouabau MC, Grolier P, Beaufrere B, Portugal H, Lairon D, Azais-Braesco V. Comparison of the postprandial plasma vitamin A response in young and older adults. J Gerontol A Biol Sci Med Sci. 1998 Mar;53(2):B133-40. doi: 10.1093/gerona/53a.2.b133. PMID 9520909
- [Background] Hubbard GP, Elia M, Holdoway A, Stratton RJ. A systematic review of compliance to oral nutritional supplements. Clin Nutr. 2012 Jun;31(3):293-312. doi: 10.1016/j.clnu.2011.11.020. Epub 2012 Jan 17. PMID 22257636
- [Background] Zhao M, Chen YH, Dong XT, Zhou J, Chen X, Wang H, Wu SX, Xia MZ, Zhang C, Xu DX. Folic acid protects against lipopolysaccharide-induced preterm delivery and intrauterine growth restriction through its anti-inflammatory effect in mice. PLoS One. 2013 Dec 6;8(12):e82713. doi: 10.1371/journal.pone.0082713. eCollection 2013. PMID 24324824
- [Background] Bazzano LA, He J, Ogden LG, Loria C, Vupputuri S, Myers L, Whelton PK. Dietary intake of folate and risk of stroke in US men and women: NHANES I Epidemiologic Follow-up Study. National Health and Nutrition Examination Survey. Stroke. 2002 May;33(5):1183-8. doi: 10.1161/01.str.0000014607.90464.88. PMID 11988588
- [Background] Bazzano LA, He J, Ogden LG, Loria CM, Vupputuri S, Myers L, Whelton PK. Fruit and vegetable intake and risk of cardiovascular disease in US adults: the first National Health and Nutrition Examination Survey Epidemiologic Follow-up Study. Am J Clin Nutr. 2002 Jul;76(1):93-9. doi: 10.1093/ajcn/76.1.93. PMID 12081821
- [Background] Varadharaj S, Kelly OJ, Khayat RN, Kumar PS, Ahmed N, Zweier JL. Role of Dietary Antioxidants in the Preservation of Vascular Function and the Modulation of Health and Disease. Front Cardiovasc Med. 2017 Nov 1;4:64. doi: 10.3389/fcvm.2017.00064. eCollection 2017. PMID 29164133
- [Background] Ji Y, Tan S, Xu Y, Chandra A, Shi C, Song B, Qin J, Gao Y. Vitamin B supplementation, homocysteine levels, and the risk of cerebrovascular disease: a meta-analysis. Neurology. 2013 Oct 8;81(15):1298-307. doi: 10.1212/WNL.0b013e3182a823cc. Epub 2013 Sep 18. PMID 24049135
- [Background] Liotet S, Cochet P, Warnet VN. [Explanation of the formation of organic deposits on soft lenses using scanning electron microscopy]. Bull Soc Ophtalmol Fr. 1983 Apr;83(4):491-3. No abstract available. French. PMID 6627576
- [Background] Ozorowski M, Wicinski M, Wrobel L, Fajkiel-Madajczyk A. Cholecalciferol supplementation lowers leptin and TMAO but increases NO and VEGF-A levels in obese vitamin D deficient patients: Is it one of the potential cardioprotective mechanisms of vitamin D? Nutr Metab (Lond). 2022 Apr 29;19(1):31. doi: 10.1186/s12986-022-00666-4. PMID 35488267
- [Background] Obeid R, Awwad HM, Kirsch SH, Waldura C, Herrmann W, Graeber S, Geisel J. Plasma trimethylamine-N-oxide following supplementation with vitamin D or D plus B vitamins. Mol Nutr Food Res. 2017 Feb;61(2). doi: 10.1002/mnfr.201600358. Epub 2016 Oct 10. PMID 27569255
- [Background] Wang X, Li X, Dong Y. Vitamin D Decreases Plasma Trimethylamine-N-oxide Level in Mice by Regulating Gut Microbiota. Biomed Res Int. 2020 Oct 5;2020:9896743. doi: 10.1155/2020/9896743. eCollection 2020. PMID 33083493
- [Background] Kalagi NA, Abbott KA, Alburikan KA, Alkofide HA, Stojanovski E, Garg ML. Modulation of Circulating Trimethylamine N-Oxide Concentrations by Dietary Supplements and Pharmacological Agents: A Systematic Review. Adv Nutr. 2019 Sep 1;10(5):876-887. doi: 10.1093/advances/nmz012. PMID 31073588
- [Background] Gatarek P, Kaluzna-Czaplinska J. Trimethylamine N-oxide (TMAO) in human health. EXCLI J. 2021 Feb 11;20:301-319. doi: 10.17179/excli2020-3239. eCollection 2021. PMID 33746664
- [Background] Masenga SK, Hamooya B, Hangoma J, Hayumbu V, Ertuglu LA, Ishimwe J, Rahman S, Saleem M, Laffer CL, Elijovich F, Kirabo A. Recent advances in modulation of cardiovascular diseases by the gut microbiota. J Hum Hypertens. 2022 Nov;36(11):952-959. doi: 10.1038/s41371-022-00698-6. Epub 2022 Apr 25. PMID 35469059
- [Background] Ercolini D, Fogliano V. Food Design To Feed the Human Gut Microbiota. J Agric Food Chem. 2018 Apr 18;66(15):3754-3758. doi: 10.1021/acs.jafc.8b00456. Epub 2018 Apr 5. PMID 29565591
- [Background] Guinane CM, Cotter PD. Role of the gut microbiota in health and chronic gastrointestinal disease: understanding a hidden metabolic organ. Therap Adv Gastroenterol. 2013 Jul;6(4):295-308. doi: 10.1177/1756283X13482996. PMID 23814609
- [Background] La Frano MR, de Moura FF, Boy E, Lonnerdal B, Burri BJ. Bioavailability of iron, zinc, and provitamin A carotenoids in biofortified staple crops. Nutr Rev. 2014 May;72(5):289-307. doi: 10.1111/nure.12108. Epub 2014 Apr 1. PMID 24689451
- [Background] Melse-Boonstra A. Bioavailability of Micronutrients From Nutrient-Dense Whole Foods: Zooming in on Dairy, Vegetables, and Fruits. Front Nutr. 2020 Jul 24;7:101. doi: 10.3389/fnut.2020.00101. eCollection 2020. PMID 32793622
- [Background] Cho CE, Taesuwan S, Malysheva OV, Bender E, Tulchinsky NF, Yan J, Sutter JL, Caudill MA. Trimethylamine-N-oxide (TMAO) response to animal source foods varies among healthy young men and is influenced by their gut microbiota composition: A randomized controlled trial. Mol Nutr Food Res. 2017 Jan;61(1). doi: 10.1002/mnfr.201600324. Epub 2016 Aug 3. PMID 27377678
- [Background] Koeth RA, Wang Z, Levison BS, Buffa JA, Org E, Sheehy BT, Britt EB, Fu X, Wu Y, Li L, Smith JD, DiDonato JA, Chen J, Li H, Wu GD, Lewis JD, Warrier M, Brown JM, Krauss RM, Tang WH, Bushman FD, Lusis AJ, Hazen SL. Intestinal microbiota metabolism of L-carnitine, a nutrient in red meat, promotes atherosclerosis. Nat Med. 2013 May;19(5):576-85. doi: 10.1038/nm.3145. Epub 2013 Apr 7. PMID 23563705
- [Background] Yang S, Li X, Yang F, Zhao R, Pan X, Liang J, Tian L, Li X, Liu L, Xing Y, Wu M. Gut Microbiota-Dependent Marker TMAO in Promoting Cardiovascular Disease: Inflammation Mechanism, Clinical Prognostic, and Potential as a Therapeutic Target. Front Pharmacol. 2019 Nov 19;10:1360. doi: 10.3389/fphar.2019.01360. eCollection 2019. PMID 31803054
- [Background] Jimenez-Torres J, Alcala-Diaz JF, Torres-Pena JD, Gutierrez-Mariscal FM, Leon-Acuna A, Gomez-Luna P, Fernandez-Gandara C, Quintana-Navarro GM, Fernandez-Garcia JC, Perez-Martinez P, Ordovas JM, Delgado-Lista J, Yubero-Serrano EM, Lopez-Miranda J. Mediterranean Diet Reduces Atherosclerosis Progression in Coronary Heart Disease: An Analysis of the CORDIOPREV Randomized Controlled Trial. Stroke. 2021 Nov;52(11):3440-3449. doi: 10.1161/STROKEAHA.120.033214. Epub 2021 Aug 10. Erratum In: Stroke. 2021 Nov;52(11):e754. doi: 10.1161/STR.0000000000000393. PMID 34372670
- [Background] Lindschinger M, Tatzber F, Schimetta W, Schmid I, Lindschinger B, Cvirn G, Fuchs N, Markolin G, Lamont E, Wonisch W. [Bioavailability of natural versus synthetic B vitamins and their effects on metabolic processes]. MMW Fortschr Med. 2020 Mar;162(Suppl 4):17-27. doi: 10.1007/s15006-020-0230-4. Epub 2020 Mar 19. German. PMID 32189314
- [Background] Zhou A, Selvanayagam JB, Hypponen E. Non-linear Mendelian randomization analyses support a role for vitamin D deficiency in cardiovascular disease risk. Eur Heart J. 2022 May 7;43(18):1731-1739. doi: 10.1093/eurheartj/ehab809. PMID 34891159
- [Background] Barbarawi M, Kheiri B, Zayed Y, Barbarawi O, Dhillon H, Swaid B, Yelangi A, Sundus S, Bachuwa G, Alkotob ML, Manson JE. Vitamin D Supplementation and Cardiovascular Disease Risks in More Than 83 000 Individuals in 21 Randomized Clinical Trials: A Meta-analysis. JAMA Cardiol. 2019 Aug 1;4(8):765-776. doi: 10.1001/jamacardio.2019.1870. PMID 31215980
- [Background] Parva NR, Tadepalli S, Singh P, Qian A, Joshi R, Kandala H, Nookala VK, Cheriyath P. Prevalence of Vitamin D Deficiency and Associated Risk Factors in the US Population (2011-2012). Cureus. 2018 Jun 5;10(6):e2741. doi: 10.7759/cureus.2741. PMID 30087817
- [Background] Orces C, Lorenzo C, Guarneros JE. The Prevalence and Determinants of Vitamin D Inadequacy among U.S. Older Adults: National Health and Nutrition Examination Survey 2007-2014. Cureus. 2019 Aug 1;11(8):e5300. doi: 10.7759/cureus.5300. PMID 31579639